CLINICAL TRIAL: NCT06820307
Title: A Phase 1, Open-label Study to Evaluate the Effect of Suzetrigine on the Pharmacokinetics of Oral Contraceptives in Healthy Female Subjects
Brief Title: Evaluation of the Effect of Suzetrigine (SUZ) on the Pharmacokinetics of Oral Contraceptives in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX24-548-019
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: SUZ with Drospirenone/Ethinyl Estradiol (DRSP/EE) (Experimental): Participants will receive a single dose of DRSP/EE on Days 1 and 20. Participants will also receive SUZ every 12 hours (q12h) from Days 7 through 25.
  Interventions: Drug: Suzetrigine; Drug: DRSP/EE
- Part B: SUZ with Norgestimate/Ethinyl Estradiol (NGM/EE) (Experimental): Participants will receive a single dose NGM/EE on Days 1 and 22. Participants will also receive SUZ every 12 hours (q12h) from Days 9 through 29.
  Interventions: Drug: Suzetrigine; Drug: NGM/EE

INTERVENTIONS:
Drug: Suzetrigine — Tablets for Oral Administration.
  Other Names: VX-548; SUZ
Drug: DRSP/EE — Combination Tablets for Oral Administration.
  Arms: Part A: SUZ with Drospirenone/Ethinyl Estradiol (DRSP/EE)
Drug: NGM/EE — Combination Tablets for Oral Administration.
  Arms: Part B: SUZ with Norgestimate/Ethinyl Estradiol (NGM/EE)

SUMMARY:
The purpose of this study is to evaluate the effect of SUZ on the pharmacokinetics of oral contraceptives.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index of 18.0 to 30.0 kilogram per meter square (Kg/m^2)
* A total body weight greater than (>) 50 kilogram (kg)
* Nonsmoker or ex-smoker for at least 12 months before screening

Key Exclusion Criteria:

* History of febrile or acute illness that has not fully resolved by 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion
* Relative contraindications to hormonal estrogen therapy that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant. This may include, but is not limited to, intolerance to hormonal contraceptives; hypertension; history of deep vein thrombosis; coronary artery disease; cardiovascular disease; systemic lupus erythematosus; migraine; history of breast or cervical cancer; cirrhosis; and history of liver cancer.

Other protocol defined Inclusion/Exclusion criteria will apply.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of DRSP and EE in the Absence and Presence of SUZ | Pre-dose up to Day 25 Post-dose
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of DRSP and EE in the Absence and Presence of SUZ | Pre-dose up to Day 25 Post-dose
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-tlast) of DRSP and EE in the Absence and Presence of SUZ | Pre-dose up to Day 25 Post-dose
Part B: Maximum Observed Plasma Concentration (Cmax) of NGM Metabolites and EE in the Absence and Presence of SUZ | Pre-dose up to Day 29 Post-dose
Part B: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of NGM Metabolites and EE in the Absence and Presence of SUZ | Pre-dose up to Day 29 Post-dose
Part B: Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-tlast) of NGM Metabolites and EE in the Absence and Presence of SUZ | Pre-dose up to Day 29 Post-dose

SECONDARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 40
Part B: Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 44

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Tempe, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing